CLINICAL TRIAL: NCT07054086
Title: Patient Derived Organoids (PDOs) to Observe the Clinical Consistency of Personalized Neoadjuvant Therapy for Resectable Esophageal Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Accurate International Biotechnology (Guangzhou) Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Tan Lijie, Chief Physician, Department of Thoracic Surgery, Shanghai Zhongshan Hospital
Other Study IDs: B2024-594R
Record Dates: First submitted 2025-05-25; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastroscopic biopsy samples; Surgical resected samples; Blood samples
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Case-group
  Interventions: Drug: Neoadjuvant Chemotherapy (NACT)

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy (NACT) — The planned regimen for neoadjuvant therapy may include one or more of the following agents:
  1. Paclitaxel Injection
  2. Albumin-bound paclitaxel Injection (Abraxane® equivalent formulation)
  3. Cisplatin Injection
  4. Carboplatin Injection
  5. Nivolumab
  6. Pembrolizumab
  7. Toripalimab
  8. Tirilibumab
  9. Camrelizumab The specific agent(s) and their combination will be selected based on the patient's clinical treatment protocol. The final regimen must be approved jointly by the principal investigator and the attending physician according to established clinical guidelines and individualized patient factors.

SUMMARY:
Study Title:

Observing Clinical Consistency of Personalized Neoadjuvant Therapy Using Patient-Derived Organoid Models (PDO) in Resectable Esophageal Squamous Cell Carcinoma

Goal:

This study aims to explore whether patient-derived organoid models (PDO)-miniature tumors grown from patients' tissue samples-can accurately predict how individuals respond to personalized pre-surgery treatments (neoadjuvant therapy) for esophageal squamous cell cancer (ESCC). The study will compare results from drug sensitivity tests performed on PDO models with actual clinical outcomes after treatment to assess consistency and potential as a predictive tool.

Main Questions Addressed:

Do PDO models accurately reflect patients' tumor characteristics and response patterns to chemotherapy/immunotherapy combinations? Can PDO drug sensitivity testing reliably predict clinical responses (treatment effectiveness) in patients receiving personalized neoadjuvant therapy?

Study Design:

This observational study will enroll patients diagnosed with resectable ESCC who undergo standard neoadjuvant therapy (chemotherapy +/- immunotherapy) before surgery. No treatments will be assigned by the study-therapy decisions remain in physicians' discretion based on standard care protocols.

Participant Procedures:

Patients will provide tissue samples (via endoscopy) used to grow PDO models and blood samples (optional) to study immune cell interactions with tumors. These samples will enable labs to test drug responses in vitro ("lab-on-a-chip" models) while patients proceed with their standard-of-care treatments and surgeries.

Key Activities:

Lab Work (non-invasive procedures post-endoscopy/surgery):

PDO models grown from tumor tissue samples (culturing process) will mimic patients' tumors in miniature (preserving biological features).

Drug sensitivity testing (chemotherapy agents like paclitaxel, platinum drugs and immunotherapies targeting PD-1/PD-L1 pathways**) will assess how tumors respond (growth inhibition rates).

Immune cell interactions (from blood samples) will model tumor-immune microenvironment responses to treatments (immunotherapy relevance).

Clinical Follow-Up:

Patients will undergo standard-of-care treatments (therapy decisions made independently) and regular monitoring post-treatment (survival follow-up every 3 months, adverse events tracked during therapy, clinical response evaluated per RECIST criteria).

Duration:

Study participation involves tissue/blood sample collection (during standard diagnostic procedures) followed by routine clinical care monitoring (treatment duration, post-surgery follow-up). Total study timeline spans March-December 2025 (1 year) with participant recruitment beginning February 2025.

Ethical Considerations:

Participants provide informed consent acknowledging optional blood sample collection (if needed) and understand study aims.

Patient identifiers removed from samples/test results ensuring confidentiality (ethical compliance).

No financial or treatment incentives-participation voluntary (patients retain autonomy) including withdrawal at any time (without affecting clinical care decisions).

Study Significance:

By bridging lab models with real-world treatment responses (PDOs validated against clinical outcomes), this research aims to develop personalized treatment strategies (precision oncology) reducing trial-and-error prescribing patterns (currently observed discrepancies in neo-adjuvant therapy responses among ESCC patients).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous cell carcinoma via endoscopic biopsy.
* Primary tumor located in the thoracic esophagus (upper third: ≤25 cm from incisors; middle third: 25-30 cm; lower third: ≥30 cm).
* Clinical staging indicates resectable ESCC based on chest/abdominal enhanced CT, neck lymph node ultrasound, PET-CT/EUS: AJCC/UICC 8th Edition clinical stage excluding T4b, ≥6 lymph node metastases, ≥3 regional lymph node stations involved/metastatic disease (M1).
* Age: 18-75 years inclusive.
* ECOG performance status score of 0 or 1, with life expectancy ≥12 months.
* Adequate organ function: WBC >4.0×10⁹/L, ANC ≥2.0×10⁹/L, platelets >100×10⁹/L, hemoglobin >90g/L; FEV1 ≥1.2L/FVC≥50%/DLCO≥50%; serum bilirubin ≤1.5×ULN; ALT/AST ≤1.5×ULN; SCr ≤120 µmol/L/Ccr ≥60 ml/min.
* Willingness and ability to provide informed consent, comply with follow-up requirements, and participate actively in drug sensitivity testing using PDO models.

Exclusion Criteria:

* Clinical staging indicates unresectable ESCC: AJCC/UICC stage T4b disease deemed inoperable by two senior thoracic surgeons; ≥6 lymph node metastases estimated clinically/regionally involving ≥3 stations with lymphadenopathy/metastasis detected via imaging (CT/PET/EUS).
* Currently receiving/was previously treated with chemotherapy/targeted therapy/radiation/or immunotherapy.
* Histopathologic diagnosis other than ESCC confirmed via biopsy (e.g., adenocarcinoma).
* History of prior malignancies except for cured cervical intraepithelial neoplasia or basal cell carcinoma limited locally.
* Autoimmune disease history; ongoing/recurrent corticosteroid/immunosuppressant use.
* Prior immunotherapy treatment; known allergy to investigational drugs; HIV/HBV(HBeAg)/HCV positivity (serum markers).
* Active interstitial lung disease/bronchiectasis; uncontrolled hypertension (SBP≥160 mmHg or DBP≥100 mmHg); cardiovascular disorders (e.g., active ischemia, arrhythmias requiring treatment).
* Pregnancy/lactation; unwillingness to use contraception during study period.
* Non-compliance with protocol requirements, psychiatric comorbidities affecting consent capacity, or concurrent participation in other clinical trials.
* Organ transplantation history (autologous bone marrow/stem cell transplant excluded).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with resectable esophageal squamous cell carcinoma (ESCC) who are enrolled from Zhongshan Hospital affiliated with Fudan University. Participants must undergo endoscopic biopsy confirmation of ESCC and preoperative clinical staging via imaging modalities (e.g., CT, PET/CT). Patients aged 18-75 years with an ECOG performance status of 0-1 and adequate organ function are eligible. The study aims to evaluate the clinical consistency between PDO-derived drug sensitivity testing and actual therapeutic responses in patients undergoing neoadjuvant therapy followed by surgical resection of ESCC tumors located in the thoracic segment (upper, middle, or lower third).
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Organoid Culture Success Metrics | before NACT accomplishment
  Assessment of the success rate in establishing patient-derived organoids (PDOs) from esophageal squamous cell carcinoma tissue samples, confirmed histologically and genomically consistent with tumor tissue.

SECONDARY OUTCOMES:
Clinical Efficacy Evaluation | 4-6 weeks after NACT complete
  Quantitative assessment of tumor response to neoadjuvant therapy using criteria from RECIST version 1.1 criteria (Complete Response [CR], Partial Response [PR], Stable Disease [SD], Progressive Disease [PD]).
Drug Sensitivity Concordance | before NACT treatment accomplishment
  Evaluation of consistency between in vitro drug sensitivity results from PDO models and clinical tumor response following neoadjuvant therapy. Key parameter: Maximum percent inhibition rate of tumor organoids exposed to programmed drug regimens (e.g., paclitaxel, pembrolizumab combinations).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT07054086/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT07054086/ICF_001.pdf